CLINICAL TRIAL: NCT02020668
Title: Phase II Study of Physiotherapy in Rheumatoid Arthritis: Randomized Single Blind Wait-list Controlled Trial
Brief Title: Efficacy of Physiotherapy on the Health and Quality of Life of the Rheumatic Patient
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Macmillan Research Group UK (Industry)
Collaborators: NMP Medical Research Institute (Other); Warwick Research Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mac/NMP 1210
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Rheumatic Arthritis
Keywords: Pain; Functional capacity; Quality of Life
MeSH Terms: conditions — Rheumatic Fever; Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiotherapy (Experimental): Physiotherapy included joint protection strategies, performance of therapeutic exercises and patient education.
  Interventions: Other: Physiotherapy
- Wait list control (Other): Wait list control received standard care and were invited to join the physiotherapy once intervention period is finished.
  Interventions: Other: Wait list control

INTERVENTIONS:
Other: Physiotherapy
  Arms: Physiotherapy
Other: Wait list control
  Arms: Wait list control

SUMMARY:
Despite leading cause of morbidity, treatment strategies for Rheumatic diseases are geared almost exclusively toward medical-pharmacological area away from offering the patient the possibility of an interdisciplinary approach to their disease.

Present study test whether treatment of physiotherapy reduces stiffness and pain inherent in rheumatic disease and improve their quality of life related to health.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* History of Rheumatoid Arthritis (RA) symptoms for less than 7 years
* Had RA by American College of Rheumatology (ACR) criteria
* ACR functional RA class I, II or III
* Hemoglobin more than 8g/dL without evidence of active bleeding
* Positive for rheumatoid factor (RF) or anti cyclic citrullinated protein
* standard conventional medicine were allowed within the approved dosage regimen

Exclusion Criteria:

* connective tissue disease
* any other alternative or complementary medicine with in last 3 months.
* corticosteroid, disease modifying medicines
* Poorly controlled diabetes, hypertension, hepatitis, cardiac disease, liver diseases, carcinoma, drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pain | Change from baseline in Numerical Scale Downie at 16 weeks

SECONDARY OUTCOMES:
Quality of Life | Change from Baseline in Short Form (SF) 36 at 16 weeks

OTHER OUTCOMES:
Functional capacity | Change from baseline in Barthel Index at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Study Director — Macmillan Research Group; Om Prakash Sharma, MBBS, Principal Investigator — Life Line Hospital, Sikar, India
Locations (1):
- Life Line Hospital, Sīkar, Rajasthan, India